CLINICAL TRIAL: NCT04755517
Title: Effectiveness of Cervical Screening in Unvaccinated, Herd Effect Protected Women - a Randomized Trial
Brief Title: Effectiveness of Cervical Screening in Unvaccinated, Herd Effect Protected Women (HPV400)
Acronym: HPV400
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other); European Union (Other); Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Tiina Eriksson, Research coordinator, Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: HPV400
Record Dates: First submitted 2021-02-04; First posted 2021-02-16 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cervical Intraepithelial Neoplasia Grade 2/3; Adenocarcinoma in Situ
Keywords: Cervical Intraepithelial Neoplasia; Neoplasms; Carcinoma in Situ; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Adenocarcinoma in situ
MeSH Terms: conditions — Adenocarcinoma in Situ; Uterine Cervical Dysplasia; Neoplasms; Carcinoma in Situ; Carcinoma; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type

STUDY DESIGN:
Who Masked: Participant
Masking Description: Frequent / Infrequent information of cytological screening results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- A1 (Active Comparator): Frequent information of screening results for cytology and/or HPV DNA at the ages of 25 (cytology only) and 28 (cytology only) vs A2
  Interventions: Other: Frequent information of cytological/ HPV DNA screening results
- A2 (No Intervention): infrequent information of cytological screening/ HPV DNA results, only at the age 28 years.
- C (Active Comparator): The third arm with at 8000 participants devoid of herd effect protection and frequent screening at ages 25 and 28 is enrolled for comparative analyses between A1 vs. C and A2 vs. C.
  Interventions: Other: Frequent information of cytological/ HPV DNA screening results

INTERVENTIONS:
Other: Frequent information of cytological/ HPV DNA screening results — All participants will be referred to pertinent diagnosis and treatment according to local standard of care (Käypä hoito 2010) should the cytological screening results (HSIL, ASC-H, AGC-FN) or three consecutive LSIL findings at repeated control visits within 3 years indicate it. The most common screening results (ASCUS, LSIL) are, however, not convened to arm A2 participants before age 28.
  All cytology and HPV DNA results results are being revealed to all trial participants at age 28 at the study end.
  Arms: A1; C

SUMMARY:
To identify: 1) Whether being informed infrequently results about screening is at least as a) safe and b) accurate as frequently obtaining all information from (the present combination of opportunistic/organized) cervical screening by comparing regimen results of two screening visits at the ages of 25 and 28 years (Arm A1) vs. results of one screening visit at the age of 28 years (Arm A2) in unvaccinated herd effect protected women. Unvaccinated, frequently screened women, who are not under herd effect protection will be controls (C).

DETAILED DESCRIPTION:
Altogether 14.000 1995-1997 born women resident in communities where herd effect against high-risk HPV infections was created with gender-neutral vaccination of birth cohorts 1992-1995 (A-communities) or not (control C-communities) in 2007-2010 with the bi-valent HPV16/18 vaccine will be invited to participate a randomized screening trial at the ages of 25 and 28 years.

Cervical samples will be analysed for HPV DNA with MGP (Modified General Primer) primer system followed by MALDITOF(matrix assisted laser desorption ionization-time of flight mass spectrometry) mass spectrometry on the SEQUENOM (translation of genomic science into solutions for molecular medicine and biomedical research) platform (HPV).

With assumed 65% and 90% participation and retain rates the trial has 80% power to show non-inferiority of the infrequent vs. the frequent screening information.

At the study-end testing the null hypotheses of no difference in the incidence of the CIN2/3 (cervical squamous intraepithelial neoplasia 2/3) end-points comparing the A1 vs. C and A2 vs. C intervention arms will be done using the Mantel-Haenszel one degree of freedom chi-square statistics.

Work Content Letters of invitation to visit cervical screening at the nearest FICAN (Comprehensive Cancer Center Finland)-Mid study site will be send to the approximately 14.000 unvaccinated women at the ages of 25 and 28 years Following informed consent cervical liquid-based cytology samples will be taken for HPV DNA and/or cytology screening at study visits.

All cytological screening results will be communicated to Arm A1 and Arm C study participants. Arm A2 participants will get the test results at the age of 28. However, results of the cytology testing indicative of colposcopy according to local standard of care and currently accepted EU (the European Union) -guidelines (Käypä Hoito 2010, Franceschi et al. 2011) will be immediately communicated to all study participants. HPV DNA results will be communicated to all study participants at the study end. Pertinent colposcopy referrals to organized health care will be made.

All study participants will be offered a possibility to give an oropharyngeal sputum sample after 30 seconds gargling of sterile physiological saline (5 ml) for HPV PCR (polymerase chain reaction) analysis.

ELIGIBILITY:
Inclusion Criteria:

* Born 1995-1997. 25 years of age residence in one of the eight community-randomized trial A communities with documented herd effect from gender-neutral vaccination or C communities devoid of the herd effect.

Exclusion Criteria:

* Immune compromising disease status (e.g. transplant recipients). HPV vaccination

Ages: 25 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 14000 (Estimated)
Dates: Start 2020-06-09 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The difference between arm A1 vs. arm C | Three years of follow up within 2020 - 2025
  No significant difference in the incidence ratios of CIN2/3 between arms A1 (participants under herd protection and frequently informed of the cytological results) vs. C (participants not under herd protection and frequently informed of the cytological findings) at the age of 28
The difference between arm A2 vs. arm C | Three years of follow up within 2020 - 2025
  No significant difference in the incidence ratios of CIN2/3 between arms A2 (participants under herd protection and frequently informed of the cytological results) vs. C (participants not under herd protection and frequently informed of the cytological findings) at the age of 28.

SECONDARY OUTCOMES:
Quality of life in infrequently vs. frequently screened unvaccinated women (RAND 36) | Three years of follow up within 2021 - 2025
  The difference between infrequently and frequently screened unvaccinated women at the age of 28 is measured using RAND 36 to measure quality of life. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Quality of life in infrequently vs. frequently screened unvaccinated women (EQ-VAS) | Three years of follow up within 2021 - 2025
  The difference between infrequently and frequently screened unvaccinated women at the age of 28 is measured using EQ-VAS a vertical visual analogue scale on which patients provide a global assessment of their health. The scale takes values between 100 (best imaginable health) and 0 (worst imaginable health).
Quality of life in infrequently vs. frequently screened unvaccinated women (CECA 10) | Three years of follow up within 2021 - 2025
  The difference between infrequently and frequently screened unvaccinated women at the age of 28 is measured using CECA 10, a Spanish acronym for the Specific Questionnaire for Condylomata Acuminata, summary scores of the emotional and sexual activity dimensions will be derived from CECA 10 scales. The CECA questionnaire includes 10 questions across 2 domains: emotional and sexual activity. CECA scores range from 0 (worst HRQL) to 100 (best HRQL)

CONTACTS AND LOCATIONS:
Overall Officials: Matti Lehtinen, MD, PhD, Principal Investigator — Tampere University
Locations (18):
- Finland (18):
  - HPV-tutkimukset, Hämeenlinna
  - HUS, Helsinki
  - HPV-tutkimukset, Iisalmi
  - HPV-tutkimukset, Joensuu
  - HPV-tutkimukset, Jyväskylä
  - Nuorisotutkimusasema, PSHP/ Tampereen yliopisto, Kemi
  - Nuorisotutkimusasema, PSHP/Tampereen yliopisto, Kotka
  - HPV-tutkimukset, Kouvola
  - Nuorisotutkimusasema, PSHP; Tampereen yliopisto, Kuopio
  - Nuorisotutkimusasema, PSHP/ Tampereen yliopisto, Lahti
  - HPV-tutkimukset, Oulu
  - HPV-tutkimukset, Pori
  - HPV-tutkimukset, Porvoo
  - Nuorisotutkimusasema, PSHP; Tampereen yliopisto, Rauma
  - HPV-tutkimukset, Sastamala
  - HPV-tutkimukset, Seinäjoki
  - Nuorisotutkimusasema; PSHP/ Tamereen yliopisto, Tampere
  - HPV-tutkimukset, Varkaus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lehtinen M, Elfstrom M, Vanska S, Dillner J. Elimination of cervical cancer by refined vaccination and screening. Int J Cancer. 2025 Feb 15;156(4):886-888. doi: 10.1002/ijc.35228. Epub 2024 Oct 25. No abstract available. PMID 39450703
- [Background] Lehtinen M, Bruni L, Elfstrom M, Gray P, Logel M, Mariz FC, Baussano I, Vanska S, Franco EL, Dillner J. Scientific approaches toward improving cervical cancer elimination strategies. Int J Cancer. 2024 May 1;154(9):1537-1548. doi: 10.1002/ijc.34839. Epub 2024 Jan 9. PMID 38196123
- [Background] Lehtinen M, Gray P, Louvanto K, Vanska S. In 30 years, gender-neutral vaccination eradicates oncogenic human papillomavirus (HPV) types while screening eliminates HPV-associated cancers. Expert Rev Vaccines. 2022 Jun;21(6):735-738. doi: 10.1080/14760584.2022.2064279. Epub 2022 Apr 15. No abstract available. PMID 35404177
- [Background] Gray P, Kann H, Pimenoff VN, Eriksson T, Luostarinen T, Vanska S, Surcel HM, Faust H, Dillner J, Lehtinen M. Human papillomavirus seroprevalence in pregnant women following gender-neutral and girls-only vaccination programs in Finland: A cross-sectional cohort analysis following a cluster randomized trial. PLoS Med. 2021 Jun 7;18(6):e1003588. doi: 10.1371/journal.pmed.1003588. eCollection 2021 Jun. PMID 34097688
- [Background] Vanska S, Luostarinen T, Baussano I, Apter D, Eriksson T, Natunen K, Nieminen P, Paavonen J, Pimenoff VN, Pukkala E, Soderlund-Strand A, Dubin G, Garnett G, Dillner J, Lehtinen M. Vaccination With Moderate Coverage Eradicates Oncogenic Human Papillomaviruses If a Gender-Neutral Strategy Is Applied. J Infect Dis. 2020 Aug 17;222(6):948-956. doi: 10.1093/infdis/jiaa099. PMID 32161969